CLINICAL TRIAL: NCT00002849
Title: Phase II Study of Dexamethasone/Alpha-Interferon in AL Amyloidosis
Brief Title: S9628 Dexamethasone Plus Interferon Alfa in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S9628; S9628 (Other: SWOG); CLB-9790 (Other: CALGB); CLB-S9628 (Other: CALGB); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Interferon-alpha; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- induction and maintenance (Experimental): dexamethasone induction followed by alpha interferon maintenance
  Interventions: Biological: recombinant interferon alfa; Drug: dexamethasone

INTERVENTIONS:
Biological: recombinant interferon alfa — first 2 years
  Other Names: alpha interferon
Drug: dexamethasone — 40 mg*/d PO 1 - 4, 9 - 12, 17-20 q 35 days for 3 cycles*
  Other Names: decadron

SUMMARY:
RATIONALE: Chemotherapy plus interferon alfa may be effective for primary systemic amyloidosis.

PURPOSE: Phase II trial to study the effectiveness of dexamethasone plus interferon alfa in treating patients who have primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate M protein and organ dysfunction responses and overall and progression-free survival in patients with primary systemic amyloidosis treated with dexamethasone/interferon alfa.
* Identify prognostic factors that may relate to response and overall survival in these patients.
* Evaluate the qualitative and quantitative toxic effects of this regimen.

OUTLINE: Patients are stratified by prior amyloidosis treatment (yes vs no).

All patients receive induction therapy with oral dexamethasone on days 1-4, 9-12, and 17-20 every 35 days for a total of 3 courses.

Maintenance therapy begins within 5-8 weeks (within 10 weeks if patients undergo stem cell harvest) of initiation of the third course of induction, as follows: oral dexamethasone for 4 days every 4 weeks; and subcutaneous interferon alfa 3 times per week. Patients who achieved less than a 50% reduction in serum M protein or urinary Bence-Jones protein and who experienced less than grade 3 toxicity during induction receive 3 additional courses of pulse dexamethasone concurrently with entry to maintenance therapy and the initiation of interferon alfa.

Combination therapy is continued until 2 years from entry; thereafter, interferon is administered alone for at least 3 years, toxicity permitting. Patients with stable disease after 5 years of therapy may discontinue interferon alfa at the discretion of the treating physician.

Patients are followed every 6 months for 2 years and yearly thereafter.

PROJECTED ACCRUAL: A total of 100 patients (50 with prior melphalan/prednisone or iododoxorubicin treatment and 50 without) will be entered over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically diagnosed primary systemic amyloidosis based on the following:

  * Deposition of fibrillary protein with Congo red positive stain or characteristic electron microscopic appearance
  * Monoclonal light chain protein (Bence-Jones protein) in serum or urine or immunohistochemical studies
  * Evidence of tissue involvement other than carpal tunnel syndrome
  * Diagnostic histologic material available for central pathology review

    * Confirmation of tissue diagnosis at all sites of organ dysfunction encouraged
* No senile, secondary, localized, dialysis-related, or familial amyloidosis
* No known therapy-related myelodysplasia

PATIENT CHARACTERISTICS:

Age:

* Adult

Performance status:

* SWOG 0-4

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No NYHA class IV status

Other:

* No uncontrolled diabetes
* No active peptic ulcer disease
* No medical condition that precludes high-dose steroids
* No second malignancy within 5 years except:
* Adequately treated nonmelanomatous skin cancer
* In situ cervical cancer
* Adequately treated stage I/II cancer in complete remission
* Not pregnant or nursing
* Effective contraception required of fertile patients
* Blood/body fluid analyses within 14 days prior to registration
* Imaging/exams for tumor measurement within 28 days prior to registration
* Other screening exams within 42 days prior to registration

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interferon alfa

Chemotherapy

* Prior melphalan allowed, but recovered from effects
* At least 4 weeks since cytotoxic therapy and recovered

Endocrine therapy

* Prior prednisone allowed, but recovered from effects
* At least 4 weeks since prior glucocorticoids
* No prior dexamethasone
* No planned or concurrent dexamethasone or other therapy for primary systemic amyloidosis

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 1996-11; Primary Completion 1998-12 (Actual); Study Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
response | 10 months
  50% or more reduction in quantitative immunoglobulin, or if the patient has light-chain disease only, a 50% or more reduction in the urine M-component (Bence-Jones protein).

CONTACTS AND LOCATIONS:
Overall Officials: Laura F. Hutchins, MD, Study Chair — University of Arkansas; Richard A. Larson, MD, Study Chair — University of Chicago
Locations (40):
- United States (40):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Dhodapkar MV, Hussein MA, Rasmussen E, Solomon A, Larson RA, Crowley JJ, Barlogie B; United States Intergroup Trial Southwest Oncology Group. Clinical efficacy of high-dose dexamethasone with maintenance dexamethasone/alpha interferon in patients with primary systemic amyloidosis: results of United States Intergroup Trial Southwest Oncology Group (SWOG) S9628. Blood. 2004 Dec 1;104(12):3520-6. doi: 10.1182/blood-2004-05-1924. Epub 2004 Aug 12. PMID 15308571
- [Result] Dhodapkar M, Jacobson J, Hussein M, et al.: High dose dexamethasone (Dex) with maintenance Dex / alpha interferon leads to improved survival in patients with primary systemic amyloidosis: results of US Intergroup Trial Southwest Oncology Group (SWOG) S9628. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2278, 2003.